CLINICAL TRIAL: NCT06791616
Title: Evaluation of Surveillance Intervals After Piecemeal Resection of Non-pedunculated Colorectal Lesions ≥20mm: SCARFACE Clinical Trial
Brief Title: Surveillance Intervals After Piecemeal Resection of Non-pedunculated Colorectal Lesions ≥20mm
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asociación Española de Gastroenterología (Other)
Collaborators: Instituto de Investigación Sanitaria y Biomédica de Alicante (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SCARFACE
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Neoplasms; Adenoma Colon; Colonic Polyps; Serrated Adenoma; Endoscopic Mucosal Resection; Non-pedunculated Lesions; Thermal Ablation; Recurrence
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps; Recurrence | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced surveillance interval (Experimental): Surveillance colonoscopies at 12 and 48 months
  Interventions: Procedure: Colonoscopy
- Standard surveillance interval (Placebo Comparator): Surveillance colonoscopies at 6, 12 and 48 months
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy — Surveillance colonoscopy

SUMMARY:
Intensive endoscopic surveillance following piecemeal resection of non-pedunculated colorectal lesions (NPCL) ≥20 mm is the current standard of care, given the high recurrence rate of these lesions (15-30%). However, most recurrences are detected at 12 months, are small and unifocal, and can be easily resected endoscopically. Furthermore, thermal margin ablation has demonstrated a reduction in recurrence rates to 5-6%, highlighting the need to optimize current surveillance protocols, which are costly, invasive, and impose a significant clinical burden.

The multicenter SCARFACE clinical trial aims to evaluate whether a reduced surveillance protocol (at 12 and 48 months) is non-inferior to the standard protocol (at 6, 12, and 48 months) in terms of recurrence rates, using a predefined non-inferiority margin. This non-inferiority design aims to determine if the reduced protocol maintains acceptable efficacy while reducing clinical workload and minimizing risks and discomfort associated with intensive follow-up.

Patients will be randomized in a 1:1 ratio into the two surveillance protocols, with an estimated sample size of 746 lesions. The primary objective is to compare the cumulative incidence of recurrence at 12 months. Secondary objectives include characterizing recurrences, assessing complications associated with endoscopic treatments and evaluating the incidence of advanced colorectal lesions. The findings of this study are expected to directly impact clinical guidelines and routine practice, optimizing resource utilization and improving patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a single non-pedunculated colorectal lesion (NPCL) ≥20 mm that has been resected piecemeal and treated with thermal ablation (using snare tip or argon plasma) at the margins as prophylaxis against recurrence, and who are awaiting the initiation of specific endoscopic follow-up.
* Complete colonoscopy with adequate or excellent bowel preparation performed within the last 6 months prior to the resection of the index lesion.
* Signed informed consent.

Exclusion Criteria:

* Resection performed using a cold snare technique due to the high risk of recurrence.
* Histology of the lesion showing malignancy: colorectal cancer with submucosal invasion, regardless of invasion depth in microns.
* Absence of information regarding the grade of dysplasia of the index lesion.
* Personal history of colorectal cancer.
* Incomplete endoscopic resection of the index lesion or any other polyps present in the patient.
* When the endoscopist performing the index colonoscopy expresses doubts about whether the resection was complete.
* Index lesion with prior attempted resection.
* Hereditary cancer syndromes (e.g., adenomatous or serrated polyposis syndromes, Lynch syndrome, etc.).
* Inflammatory bowel disease.
* Severe comorbidities with reduced life expectancy.
* Pregnancy.
* Ongoing cytotoxic treatment or radiotherapy for a malignant disease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 746 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of recurrence/residual tissue | 12 months

SECONDARY OUTCOMES:
To compare the cumulative incidence of recurrence/residual tissue | 48 months
To describe the characteristics of recurrences | 48 months
To determine the complete endoscopic resection rate in patients who have experienced recurrence. | 48 months
To analyze the incidence of complications arising from the endoscopic treatment of recurrences. | 48 months
To determine the proportion of patients requiring surgery to treat recurrence or complications associated with it. | 48 months
To assess the incidence of advanced colonic lesions or colorectal cancer | 12 months
To assess the incidence of advanced colonic lesions or colorectal cancer | 48 months

IPD SHARING:
Plan to Share IPD: No